CLINICAL TRIAL: NCT02878018
Title: Cohort Study on Traditional Chinese Medicine Diagnosis and Treatment of Children With Henoch-Schonlein Purpura Nephritis
Acronym: CSTCMDTCHSPN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: First Hospital of China Medical University (Other); Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Zhang Jun, Professor, Liaoning University of Traditional Chinese Medicine
Other Study IDs: ZJ16813
Record Dates: First submitted 2016-08-17; First posted 2016-08-25 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Henoch-Schonlein Purpura Nephritis
Keywords: Cohort Study; Children; Henoch-Schonlein Purpura Nephritis; Traditional Chinese Medicine
MeSH Terms: interventions — Dipeptidyl-Peptidases and Tripeptidyl-Peptidases; Adrenal Cortex Hormones; Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — We will retain the blood of each patient to do some research of lncRNA with patients'permission.Try to find some relationship between lncRNA and HSPN disease.We also retain the urine and coated tongue to establish the biospecimen repository for our patients.When they grow up,these spicimens may help them to understand their bodies more correctly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCM intervention: Participants with HSPN of the Heat-Toxin type will take the Qi-Ji Shen-Kang formula. HSPN patients of the Wet-Heat type will take the Zhu-Bai formula. Those of Qi-Deficiency with Blood-Stasis type will take the Yu-Shen formula.
  Interventions: Drug: Qi-Ji Shen-Kang formula; Zhu-Bai formula; Yu-Shen formula
- WM conventional intervention: The WM conventional intervention, recommended by the Chinese Medical Association's (CMA) Scientific Statement, includes angiotensin-converting enzyme (ACE) inhibitor, adrenergic receptor binder (ARB), adrenal cortical hormone, Tripterygium wilfordii polyglycosidium and an immunosuppressant.
  Interventions: Drug: angiotensin-converting enzyme (ACE) inhibitor; adrenergic receptor binder (ARB); adrenal cortical hormone; Tripterygium wilfordii polyglycosidium; immunosuppressant

INTERVENTIONS:
Drug: Qi-Ji Shen-Kang formula; Zhu-Bai formula; Yu-Shen formula — Qi-Ji Shen-Kang formula:15g of field thistle,10g of common edelweiss herb,10g of spreading hedyotis herb,10g ofYunnan manyleaf Paris rhizome,10g of hairyvein agrimonia herb,10g of the root bark of the tree peony,15g of root of red rooted salvia, and 15g ofmembranous mikvetch root.Zhu-Bai formula:10g of glabrous greenbrier rhizome,5g of Chinese atractylodes rhizome,10g of amur corktree bark,10g of common edelweiss her),10g of field thistle,10g of lalang grass rhizome,10g of garden burnet root,5g of longbract cattail pollen,5g of rehmanniae radix, and 5g of Chinese angelica root.Yu-Shen formula:15g of membranous mikvetch root,10g of heterophylla falsestarwort root,10g of field thistle,10g of cogongrass rhizome,10g of spreading hedyotis herb,10g of root of red rooted salvia,10g of fresh root of rehmannia,10g of Asian puccoon,10g of wormwoodlike motherwort herb,10g of common cockscomb inflorescence,10g of gordon euyale,10g of root bark of the tree peony, and 5g of licorice root.
  Groups: TCM intervention
Drug: angiotensin-converting enzyme (ACE) inhibitor; adrenergic receptor binder (ARB); adrenal cortical hormone; Tripterygium wilfordii polyglycosidium; immunosuppressant — prednisone at a dose of 1-1.5 mg/(kg·d) and Tripterygium wilfordii polyglycosidium at a dose of 1 mg/(kg·d). For each patient, the specific Western medicines used and their doses may be adjusted at the discretion of his or her physician, but the classes cannot be changed.
  Groups: WM conventional intervention

SUMMARY:
Henoch-Schonlein purpura nephritis(HSPN) is one of the most common secondary glomerulonephritis in children. A large, prospective, multicenter cohort study is being conducted in three institutions. Eligible Henoch-Schönlein purpura nephritis children will be classified as the experimental group (n=300) and the control group (n=300) based on the interventions they receive. Patients taking Chinese herbal formula will be in the experimental group, and those taking Western medicine will be in the control group. The entire study will last 60 weeks, including a 12-week observation period and a followup at 12 months.

DETAILED DESCRIPTION:
Background: Henoch-Schönlein purpura nephritis involves the renal impairment of Henoch-Schönlein purpura and can easily relapse into life-threatening late nephropathy in severe cases. Although there is a lack of validated evidence for its effectiveness, traditional Chinese medicine is the most commonly used method in China to treat Henoch-Schönlein purpura nephritis. We report the protocol of a prospective cohort trial using traditional Chinese medicine to investigate the effectiveness, safety and advantages for children with Henoch-Schönlein purpura nephritis.

Methods/Design: A large, prospective, multicenter cohort study is being conducted in three institutions. Eligible Henoch-Schönlein purpura nephritis children will be classified as the experimental group (n=300) and the control group (n=300) based on the interventions they receive. Patients taking Chinese herbal formula will be in the experimental group, and those taking Western medicine will be in the control group. The entire study will last 60 weeks, including a 12-week observation period and a followup at 12 months. Seven visits will be scheduled for each participant with visits in week 0, week 2, week 4, week 6, week 8, week 10 and week 12. The primary outcomes include the remission rate and the recurrence rate. The secondary outcomes include the urine erythrocyte effectiveness, the urine protein effectiveness, the hormone usage rate, the immunosuppressant usage rate, and the incidence rate of renal failure. Safety outcomes and any adverse reactions will be recorded during the study.

Discussion: This study will determine whether the Chinese herbal formula is helpful for treating Henoch-Schönlein purpura nephritis in children. The findings will provide a basis for further confirmatory studies.

ELIGIBILITY:
Inclusion criteria

1. A diagnosis of HSPN as well as three major constitution types (Heat-Toxin, Wet-Heat, Qi-Deficiency with Blood-Stasis) according to WM and TCM.
2. Age: 5 to 18 years old (including 5 and 18 year-olds).
3. The clinical classification of HSPN includes isolated hematuria, insolated proteinuria, hematuria with proteinuria, and acute glomerulonephritis.
4. The ability to provide detailed connection and complete a followup.
5. The ability to understand and sign a written informed consent.

Exclusion criteria

1. HSPN with renal insufficiency.
2. A clinical classification of HSPN that includes nephritic syndrome, rapidly progressive glomerulonephritis and chronic glomerulonephritis.
3. Suffering from serious complications, such as respiratory, digestive, hematological or liver diseases.
4. Tumor, infectious diseases, or mental disorders.
5. Allergic to TCM use.
6. No prescribed medication, poor compliance, or incomplete data affecting the efficacy and safety of these judgments.
7. A history of another clinical trial in the previous 2 weeks.
8. No consent form signed.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with purpura nephritis who are treated in Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shengjing Hospital of China Medical University and The First Hospital of China Medical University will be regarded as the objects of study.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-09; Primary Completion 2019-03 (Actual); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Urine protein | 2 weeks
  1. Recovery:Urine protein(-).
  2. Marked effect:Urine protein reduces by 2'+'.
  3. Effective：Urine protein reduces by 1'+'.
  4. Ineffective：Urine protein has no changes.
24-hour urinary protein excretion | 2 weeks
  1. Recovery:24-hour urinary protein excretion is normal.
  2. Marked effect:24-hour urinary protein excretion reduction is larger than 50%.
  3. Effective：24-hour urinary protein excretion reduction is smaller than 50%.
  4. Ineffective：24-hour urinary protein excretion has no changes.
Urine erythrocyte | 2 weeks
  1. Recovery:Urine erythrocyte is normal.
  2. Marked effect:Urine erythrocyte reduction is larger than 50%.
  3. Effective:Urine erythrocyte reduction is smaller than 50%.
  4. Ineffective；Urine erythrocyte has no changes.
Creatinine clearance rate and Serum creatinine | 1 year
  Diagnostic criteria of chronic renal failure:
  1. Creatinine clearance rate<80ml/min;
  2. Serum creatinine>133μmol/L;
  3. The patient who have a history of chronic kidney diseases or systemic diseases involving kidney.

SECONDARY OUTCOMES:
Number of patients with hormone therapy | 3 months
  Hormone utilized rate=Number of patients with hormone therapy/The total number of patients
Number of patients with immunosuppressant therapy | 3 months
  Immunosuppressant utilized rate=Number of patients with immunosuppressant therapy/The total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: jun zhang, master, Study Chair — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; jing lv, master, Study Director — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; shaoqing zhang, doctor, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; guanqi yang, doctor, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; shuang pang, doctor, Principal Investigator — Affiliated Hospital of Liaoning University of Traditional Chinese Medicine; binyu wu, master, Principal Investigator — Shengjing Hospital; yaoguo zhang, master, Principal Investigator — First Hospital of China Medical University
Locations (1):
- Zhang Jun, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
The Central Database of Clinical Evaluation of China Academy of Chinese Medicine Science

REFERENCES:
- [Derived] Zhang J, Lv J, Pang S, Bai X, Yuan F, Wu Y, Jiang H, Yang G, Zhang S. Chinese herbal medicine for the treatment of Henoch-Schonlein purpura nephritis in children: A prospective cohort study protocol. Medicine (Baltimore). 2018 Jun;97(24):e11064. doi: 10.1097/MD.0000000000011064. PMID 29901610